CLINICAL TRIAL: NCT03350698
Title: Occupational Exposure to Human Papilloma Virus (HPV) and Prophylactic Vaccination (Version IV Dated 24Oct2017)
Brief Title: Occupational Exposure to Human Papilloma Virus (HPV) and Prophylactic Vaccination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Craig Derkay M.D., Professor, Eastern Virginia Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-09-FB-0176
Record Dates: First submitted 2017-11-10; First posted 2017-11-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Papillomavirus Vaccines
Keywords: Human papilloma virus

STUDY DESIGN:
Intervention Model Description: Prospective Single-Subject Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- active drug (Experimental): Human Papilloma virus ,Gardasil, 9 valent vaccine
  Interventions: Biological: Gardasil-9

INTERVENTIONS:
Biological: Gardasil-9 — 3 vaccine series

SUMMARY:
Currently there are no standards for healthcare worker vaccination with the HPV, Gardasil-9 vaccine. For health care workers, the CDC only recommends for vaccination against hepatitis B, influenza virus, Measles, Mumps and Rubella (MMR), Chickenpox (Varicella), Tetanus, Diptheria, and Pertussis (Tdap), and meninogococcal infections6

DETAILED DESCRIPTION:
Initial antibody titers will be measured immediately prior to initial vaccination (month 0). This will entail a blood-draw sample (less than 1 teaspoon) that will be sent to FOCUS labs for evaluation. This will be paid for by funding received from Merck.

The three-dose vaccination schedule will be followed with injections at month 0, 2, and 6. Gardasil 9 dosing will be per the recommended and approved labeled guidelines. Post-vaccination titers would be measured at month 7, which is in alignment with the methods of previous studies. This will entail a blood-draw sample (less than 1 teaspoon) that will be sent to FOCUS labs for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* • Actively practicing attending surgeon in the field of Otolaryngology, General Surgery, Urology, or Obstetrics-Gynecology employed by EVMS or credentialed by CHKD and/or SNGH.

or

• Current residents of EVMS Otolaryngology, General Surgery, Urology, or Obstetrics-Gynecology programs

Exclusion Criteria:

* • Age 26 or younger

  * Age over 69
  * Hypersensitivity to vaccine component
  * History of severe allergic or hypersensitivity reactions to yeast
  * History of previous HPV vaccination with 9 valent vaccine
  * Pregnant
  * Moderate or severe acute illness

Ages: 27 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
# of participants with elevated HPV antibody titers from baseline to 7 months | baseline and 7 months
  baseline change at 7 months post vaccine series. The antibody titer laboratory test will be used to record the levels

CONTACTS AND LOCATIONS:
Overall Officials: Craig H Derkay, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- EVMS Otolaryngology, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marur S, D'Souza G, Westra WH, Forastiere AA. HPV-associated head and neck cancer: a virus-related cancer epidemic. Lancet Oncol. 2010 Aug;11(8):781-9. doi: 10.1016/S1470-2045(10)70017-6. Epub 2010 May 5. PMID 20451455
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Dickens P, Srivastava G, Loke SL, Larkin S. Human papillomavirus 6, 11, and 16 in laryngeal papillomas. J Pathol. 1991 Nov;165(3):243-6. doi: 10.1002/path.1711650308. PMID 1662265
- [Background] Stransky N, Egloff AM, Tward AD, Kostic AD, Cibulskis K, Sivachenko A, Kryukov GV, Lawrence MS, Sougnez C, McKenna A, Shefler E, Ramos AH, Stojanov P, Carter SL, Voet D, Cortes ML, Auclair D, Berger MF, Saksena G, Guiducci C, Onofrio RC, Parkin M, Romkes M, Weissfeld JL, Seethala RR, Wang L, Rangel-Escareno C, Fernandez-Lopez JC, Hidalgo-Miranda A, Melendez-Zajgla J, Winckler W, Ardlie K, Gabriel SB, Meyerson M, Lander ES, Getz G, Golub TR, Garraway LA, Grandis JR. The mutational landscape of head and neck squamous cell carcinoma. Science. 2011 Aug 26;333(6046):1157-60. doi: 10.1126/science.1208130. Epub 2011 Jul 28. PMID 21798893
- [Background] Hallmo P, Naess O. Laryngeal papillomatosis with human papillomavirus DNA contracted by a laser surgeon. Eur Arch Otorhinolaryngol. 1991;248(7):425-7. doi: 10.1007/BF01463570. PMID 1660719
- [Background] Calero L, Brusis T. [Laryngeal papillomatosis - first recognition in Germany as an occupational disease in an operating room nurse]. Laryngorhinootologie. 2003 Nov;82(11):790-3. doi: 10.1055/s-2003-44546. German. PMID 14634897
- [Background] Makiyama K, Hirai R, Matsuzaki H. Gardasil Vaccination for Recurrent Laryngeal Papillomatosis in Adult Men: First Report: Changes in HPV Antibody Titer. J Voice. 2017 Jan;31(1):104-106. doi: 10.1016/j.jvoice.2016.01.008. Epub 2016 Apr 8. PMID 27068425
- [Background] Einstein MH, Takacs P, Chatterjee A, Sperling RS, Chakhtoura N, Blatter MM, Lalezari J, David MP, Lin L, Struyf F, Dubin G; HPV-010 Study Group. Comparison of long-term immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and HPV-6/11/16/18 vaccine in healthy women aged 18-45 years: end-of-study analysis of a Phase III randomized trial. Hum Vaccin Immunother. 2014;10(12):3435-45. doi: 10.4161/hv.36121. PMID 25483701
- [Background] Sehulster L, Chinn RY; CDC; HICPAC. Guidelines for environmental infection control in health-care facilities. Recommendations of CDC and the Healthcare Infection Control Practices Advisory Committee (HICPAC). MMWR Recomm Rep. 2003 Jun 6;52(RR-10):1-42. PMID 12836624
- [Background] Ilmarinen T, Auvinen E, Hiltunen-Back E, Ranki A, Aaltonen LM, Pitkaranta A. Transmission of human papillomavirus DNA from patient to surgical masks, gloves and oral mucosa of medical personnel during treatment of laryngeal papillomas and genital warts. Eur Arch Otorhinolaryngol. 2012 Nov;269(11):2367-71. doi: 10.1007/s00405-012-2049-9. Epub 2012 May 16. PMID 22588197
- [Background] Garden JM, O'Banion MK, Bakus AD, Olson C. Viral disease transmitted by laser-generated plume (aerosol). Arch Dermatol. 2002 Oct;138(10):1303-7. doi: 10.1001/archderm.138.10.1303. PMID 12374535
- See also: recommended vaccines for healthcare workers — http://www.cdc.gov/vaccines/adults/rec-vac/hcw.html